CLINICAL TRIAL: NCT04052490
Title: Evaluation Of Zirconia Crowns Restoring Endodontically Treated Posterior Teeth With Two Finish Line Designs And Occlusal Reduction Schemes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Samir Fathy El-Ashkar, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEBC-CU-2019915
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Gingival Inflammation
Keywords: Zirconia,; occlusal scheme,; endodontically treated teeth,; finishline designs.
MeSH Terms: conditions — Gingivitis; Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- flat occlusal reduction with feather edge finish (Experimental)
  Interventions: Other: Abutment with flat occlusal reduction with feather edge finish
- flat occlusal reduction with shoulder finish line (Experimental)
  Interventions: Other: Abutment with flat occlusal reduction with feather edge finish
- planar occlusal reduction with shoulder finish line (No Intervention)

INTERVENTIONS:
Other: Abutment with flat occlusal reduction with feather edge finish — Non vital teeth require a full coverage restoration to withstand the functional stresses and prevent any further destruction of tooth/crown complex. The zirconia all-ceramic crowns yield a high flexure strength and are used as an esthetic alternative to ceramo-metallic crowns. Several studies linked the effect of preparation designs to the survival of the restoration. Others, studied the effect of the finish line geometries as deep chamfer and shoulder on the marginal integrity of restorations. The feather edge finish line is used with zirconia crowns with limited data regarding its success. However, there is no presented research dealing with the effect of finishing line designs in combination with different occlusal reduction schemes on the marginal fit of full contour zirconia crowns.
  Other Names: Experimental: Abutment with flat occlusal reduction with shoulder finish line
  Arms: flat occlusal reduction with feather edge finish; flat occlusal reduction with shoulder finish line

SUMMARY:
The aim of this study is to evaluate the clinical performance of two finish line designs (feather edge and rounded shoulder) in relation with two occlusal designs (flat and planar) in endodontically treated teeth restored with zirconia crowns.

DETAILED DESCRIPTION:
Several studies have been investigating the effect of preparation design and its relation to the marginal adaptation. Habib et al 2014 compared the accuracy of marginal and internal adaptation of zirconia copings fabricated on anatomic (A), semi-anatomic (SA) and non-anatomic (NA) occlusal surface preparations. The internal & marginal fit were measured under electron microscope at 9 standardized areas .The anatomical occlusal preparation had better marginal and internal adaptation of Zr copings. Lima et al 2018 studied the influence of two different occlusal preparation designs on the marginal adaptation of CAD-CAM onlay restorations. The conventional anatomical occlusal preparation with a 1.2-mm modified shoulder finish line extending on the buccal surface and modified preparation flat cuspal reduction without shoulder finish line. The results showed that the conventional anatomical occlusal preparation had significantly better marginal adaptation than that of the flat cuspal preparation. Succeeding these studies, it was of interest to investigate whether or not the occlusal scheme could influence the marginal accuracy of the CAD/CAM crowns fabricated with Zirconia ceramic material.

Studies correlating between the finish line design and occlusal scheme in literature are scarce, with little evidence regarding their effect on precision fit properties of restorations. Abdullah et al 2017 evaluated the effect of using different finishing line designs with different occlusal surface reduction schemes on the vertical marginal fit of full contour CAD/CAM zirconia crown restorations. They found a direct correlation between both the finish line geometry and the occlusal design. In recent literature, the use of feather edge finish line with all ceramic restorations is a point of conflict. Fuzzi et al 2017 studied the nanoleakage and internal adaptations of lithium disilicate and zirconia crowns with featheredge finish lines. They recommended only zirconia with this finish line configuration due to its high fracture resistance when used in thin sections. Thus, the current study was conducted to examine this finish line effect on the marginal precision fit. Our hypothesis is there will be no difference in the clinical performance between the flat occlusal scheme with feather edge or rounded shoulder finish line and the planar occlusal scheme with rounded shoulder finish line configuration.

The rationale for carrying out the trial:

The influence of different tooth preparation designs can affect the success of the full coverage restorations. Still, there is no available research dealing with the effect of finishing line designs in combination with different occlusal reduction schemes on the marginal fit of full contour zirconia crowns.

ELIGIBILITY:
Inclusion Criteria:

* From 21-50 years old, be able to read and sign the informed consent document.
* Have no active periodontal or periapical diseases.
* Psychologically and physically able to withstand conventional dental procedures.
* Maintenance of good oral hygiene.
* Patients with teeth problems indicated for single posterior crowns:
* Badly decayed teeth
* Sufficient occluso-gingival tooth height
* Endodontically treated teeth
* No tooth mobility or grade 1 can be accepted.
* No furcation involvement.
* Able to return for follow-up examinations and evaluation.

Exclusion Criteria:

* Patients with defective root canal treatment
* Patient with active resistant periodontal diseases
* Patients with poor oral hygiene and uncooperative patients
* Pregnant women
* Patients in the growth stage with partially erupted teeth
* Psychiatric problems or unrealistic expectations
* Lack of opposing dentition in the area of interest
* Patients with bruxism.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
clinical performance in terms of the marginal adaptation of the groups | One-Year
  examination will follow the USPHS criteria.

SECONDARY OUTCOMES:
the fracture of the restoration | One-year
  examination will follow the USPHS criteria.
marginal discoloration | One-year
  examination will follow the USPHS criteria.
secondary caries | One-year
  examination will follow the USPHS criteria.
gingival response | One-year
  examination will follow the gingival index criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo university, Cairo, Manial, Egypt